CLINICAL TRIAL: NCT00003486
Title: Phase II Study of Antineoplastons A10 and AS2-1 Capsules in Patients With Adenocarcinoma of the Colon
Brief Title: Antineoplaston Therapy in Treating Patients With Colon Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BC-CO-3; CDR0000066524 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Stage IV Colon Cancer; Recurrent Colon Cancer; Adenocarcinoma of the Colon
MeSH Terms: conditions — Colonic Neoplasms | interventions — antineoplaston A10; antineoplaston AS 2-1; Biological Therapy; Complementary Therapies

INTERVENTIONS:
Drug: antineoplaston A10
Drug: antineoplaston AS2-1
Procedure: alternative product therapy
Procedure: biological therapy
Procedure: biologically based therapies
Procedure: cancer prevention intervention
Procedure: complementary and alternative therapy
Procedure: differentiation therapy

SUMMARY:
RATIONALE: Antineoplastons are naturally occurring substances that may also be made in the laboratory. Antineoplastons may inhibit the growth of cancer cells.

PURPOSE: This phase II trial is studying how well antineoplaston therapy works in treating patients with colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of antineoplastons A10 and AS2-1 in patients with adenocarcinoma of the colon by determining the proportion of patients who experience an objective tumor response.
* Evaluate the adverse effects of and tolerance to this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive gradually escalating doses of oral antineoplaston A10 and oral antineoplaston AS2-1 6-7 times a day. If the patient has not achieved a partial or complete response after 3-4 months of treatment, the investigator may discontinue treatment. Patients with stable disease may continue to receive treatment until disease progression or unacceptable toxicity is observed.

Tumors are measured every 4 months during the first 2 years, then every 6 months during years 3 and 4, and yearly during years 5 and 6.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon that is unlikely to respond to existing therapy and for which no curative therapy exists
* Measurable disease by MRI or CT scan
* Metastatic or unresectable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No renal failure

Cardiovascular:

* No chronic heart failure
* No uncontrolled hypertension

Pulmonary:

* No serious lung disease, such as chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No active infection
* No serious malabsorption syndromes
* No other serious concurrent disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered (patients with multiple tumors may be admitted earlier)

Surgery:

* No prior extensive stomach or intestinal surgery

Other:

* Prior cytodifferentiating agent allowed
* No prior antineoplaston therapy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Study Chair — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States